CLINICAL TRIAL: NCT05470855
Title: A Clinical Trial to Evaluate Protective Effect, Safety and Immunogenicity of Live Attenuated Varicella Vaccine in Children Aged 1-12 Years
Brief Title: Protective Effect, Safety and Immunogenicity of Live Attenuated Varicella Vaccine in Anhui Province
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-VAR-MA4003-AH
Record Dates: First submitted 2022-07-12; First posted 2022-07-22 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-07

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group in Protective effect study (Experimental): 22500 subjects including 7500 subjects aged 1-3 years with no history of varicella vaccination,7500 subjects aged 4-6 years with a history of 1 dose of varicella vaccine,7500 subjects aged 7-12 years with a history of 1 dose of varicella vaccine will receive one dose of varicella vaccine.
  Interventions: Biological: Live attenuated varicella vaccine
- Control Group in Protective effect study (No Intervention): 22500 subjects including 7500 subjects aged 1-3 years with no history of varicella vaccination,7500 subjects aged 4-6 years with a history of 1 dose of varicella vaccine,7500 subjects aged 7-12 years with a history of 1 dose of varicella vaccine.
- Safety group (Experimental): 30000 subjects from study 1 will be enrolled to conduct safety observation study,all adverse events of all subjects will be collected.
  Interventions: Biological: Live attenuated varicella vaccine
- Etiological study group (Experimental): Herpes fluid collected from varicella cases in study 1 will be used to conduct etiological study on the pathogenic strains of varicella cases.
  Interventions: Biological: Live attenuated varicella vaccine

INTERVENTIONS:
Biological: Live attenuated varicella vaccine — The live attenuated varicella vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd. Live attenuated varicella-virus in 0.5 mL injection water with sucrose,sodium glutamate,sodium chloride,potassium chloride, sodium dihydrogen phosphate, potassium dihydrogen phosphate per injection.The routine of administration is intramuscular injection into deltoid region of the lateral upper arm.
  Arms: Etiological study group; Experimental Group in Protective effect study; Safety group

SUMMARY:
This is Phase 4 clinical trial of live attenuated varicella vaccines manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd .The purpose of this study is to evaluate the protective effect of varicella vaccine in children aged 1-12 years and the correlation between varicella antibody and protective effect,to evaluate the immunogenicity and safety of varicella vaccine in children aged 1-12 years.

DETAILED DESCRIPTION:
This study is Phase Ⅳ clinical trial.The experimental vaccine manufactured by Sinovac(Dalian) Vaccine Technology Co., Ltd.This clinical trial consists of four parts,and A total of 45400 subjects will be enrolled.

Study 1,45000 subjects including 15000 subjects aged 1-3 years with no history of varicella vaccination ,15000 subjects aged 4-6 years with a history of 1 dose of varicella vaccine,15000 subjects aged 7-12 years with a history of 1 dose of varicella vaccine will be enrolled to evaluate protective effect of varicella vaccine. There will be 7500 subjects in the experimental group and 7500 in the control group in each age group.And subjects who voluntarily receive varicella vaccine will be included in the experimental group and other subjects will be included in the control group.All subjects in the experimental group will receive one dose of varicella vaccine.

Study 2,400 healthy children including 100 subjects aged 1-3 years with no history of varicella ,150 subjects aged 4-6 years(50 children with no history of varicella vaccination and 100 children with a history of one dose of varicella vaccine),150 subjects aged 7-12 years (50 children with no history of varicella vaccination and 100 children with a history of one dose of varicella vaccine),each subject will receive one or two doses (0,3 months) of varicella vaccine.

Study 3,30000 subjects from study 1 will be enrolled to conduct safety observation study,all adverse events of all subjects will be collected.

Study 4,Herpes fluid collected from study 1 varicella cases will be used to conduct etiological study on the pathogenic strains of varicella cases.

ELIGIBILITY:
Study 1: Inclusion criteria for a protective effect study of varicella vaccine:

* Healthy children aged 1-12 years without a history of varicella;
* The subjects and/or guardians can understand and voluntarily sign the informed consent form (For subjects aged 8 years and above, both subjects and guardians need to sign the informed consent form);

Study 2: Inclusion criteria for immunogenicity and safety evaluation of varicella vaccine:

* Healthy children aged 1-12 years without a history of varicella;
* The subjects and/or guardians can understand and voluntarily sign the informed consent form (For subjects aged 8 years and above, both subjects and guardians need to sign the informed consent form);
* The subjects and their guardians voluntarily participate in the study and are able to follow all study procedures;
* Proven legal identity.

Study 3: Inclusion criteria for safety evaluation of mass vaccination of varicella vaccine :

* Healthy children aged 1-12 years without a history of varicella;
* The subjects and/or guardians can understand and voluntarily sign the informed consent form (For subjects aged 8 years and above, both subjects and guardians need to sign the informed consent form);
* The subjects and their guardians voluntarily participate in the study and are able to follow all study procedures;
* Proven legal identity;
* Subjects'guardians can fill in adverse events using mobile apps;

Study 4: Inclusion criteria for etiological study on the pathogenic strains of varicella cases:

* Varicella cases among study 1 enrolled subjects who signed informed consent for biological samples collection.

Exclusion Criteria:

* Received two doses of varicella vaccine from other manufacturers(applied to study 1 exclusion criteria);
* Received two doses of varicella vaccine;
* History of severe allergic reactions to vaccines (e.g.acute anaphylaxis, angioneurotic edema, dyspnea, etc.);
* Any confirmed or suspected immunodeficiency disease, including human immunodeficiency virus (HIV) infection;
* Axillary temperature >37.0°C;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 28 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45400 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-02-10 (Estimated)

PRIMARY OUTCOMES:
The incidence density | 42 days after vaccination
  The incidence density will be calculated by the number of confirmed cases of varicella at 42 days after vaccination.
The protection rate | 42 days after vaccination
  The protection rate will be calculated by the number of confirmed cases of varicella at 42 days after vaccination.

SECONDARY OUTCOMES:
GMT of varicella antibody | 42 days after varicella vaccination
  GMT of varicella antibody at 42 days after varicella vaccination.
GMI of varicella antibody | 42 days after varicella vaccination
  GMI of varicella antibody at 42 days after varicella vaccination.
Positive rates of varicella antibody | 42 days after varicella vaccination
  Positive rate of varicella antibody at 42 days after varicella vaccination.
Immunogenicity index-GMT of varicella antibody | 4 months after varicella vaccination
  GMT of varicella antibody at 4 months after varicella vaccination.
Immunogenicity index-GMI of varicella antibody | 4 months after varicella vaccination
  GMI of varicella antibody at 4 months after varicella vaccination.
Immunogenicity index- positive rates | 4 months after varicella vaccination
  Positive rates of varicella antibody at 4 months after varicella vaccination.
The incidence of adverse events, serious adverse events and adverse reactions | 14 days after varicella vaccination
  The incidence of adverse events, serious adverse events and adverse reactions at 14 days after varicella vaccination.
Incidence of adverse events, serious adverse events and adverse reactions | 42 days after varicella vaccination.
  The incidence of adverse events, serious adverse events and adverse reactions at 42 days after varicella vaccination.
Safety index-Incidence of adverse events, serious adverse events and adverse reactions | 3 months after varicella vaccination
  The incidence of adverse events, serious adverse events and adverse reactions in 3 months after varicella vaccination.
Safety index-incidence of adverse events, serious adverse events and adverse reactions | 6 months after varicella vaccination
  The incidence of adverse events, serious adverse events and adverse reactions in 6 months after varicella vaccination.
Safety index- incidence of adverse events, serious adverse events and adverse reactions | 9 months after varicella vaccination
  The incidence of adverse events, serious adverse events and adverse reactions in 9 months after varicella vaccination.
The incidence of adverse events, serious adverse events and adverse reactions | 12 months after varicella vaccination
  The incidence of adverse events, serious adverse events and adverse reactions in 12 months after varicella vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Jihai Tang, Master, Principal Investigator — Anhui Provincial Center for Disease Prevention and Control
Locations (5):
- China (5):
  - Susong County Center for Disease Control and Prevention, Anqing, Anhui
  - Laian Center for Disease Control and Prevention, Chuzhou, Anhui
  - Funan County Center for Disease Control and Prevention, Fuyang, Anhui
  - Huoqiu County Center for Disease Control and Prevention, Liu‘an, Anhui
  - Ningguo Center for Disease Control and Prevention, Xuancheng, Anhui